CLINICAL TRIAL: NCT01564953
Title: Serum Magnesium and Nit Vitamin D is Associated With Better QoL in COPD: A Cross-sectional Study
Brief Title: Magnesium is Associated With QoL in COPD: A Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M-20110280
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2013-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: vitamin D; calcium; magnesium; COPD; QoL
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples:
  p-creatinine p-potassium p-sodium p-albumine p-phosphate p-magnesium p-calcium-ion p-parathyrine p-25-hydroxy-vitamin D2 + D3
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to investigate the associations between serum concentrations of vitamin D, Magnesium and Calcium in Chronic obstructive pulmonary disease patients and the potential impact of these parameters on lung function and quality of life.

DETAILED DESCRIPTION:
Attention is enhancing worldwide on the increasing tendency of insufficient 25-hydroxyvitamin D serum levels. New insights into the role of vitamin D and distribution of its receptors in the human body have been revealed. Presumably, this entails implications concerning disease and treatment that go far beyond the well-known field of bone-metabolism.

Vitamin D deficiency is common in patients with chronic obstructive pulmonary disease (COPD), and reductions in vitamin D serum levels have formerly been perceived as a consequence rather than a cause of COPD.

Yet, there is a lack of consensus concerning the role of vitamin D on the decreasing lung function in COPD.

Some trials have revealed a high degree of co-variation between the grade of airway obstruction, intake of vitamin D and reduction of serum-vitamin D. Other claim that vitamin D appears to be capable of inhibiting pulmonary inflammatory responses.

Vitamin D interacts with calcium and magnesium and this subtle balance might be highly relevant in the progression of inflammatory diseases like COPD. Presumably, Mg inhibits contraction and relaxes smooth muscles in airways due to blocking of calcium-ion-flux across the cell membrane.

The aim of this study is to investigate the status of vitamin D, magnesium and calcium in COPD, and to study the relationship and impact of vitamin D, magnesium and calcium in COPD-patients.

The hypothesis of this study is that COPD-patients with vitamin D-, magnesium- and calcium supplement have a better lung function and quality of life, than those who have vitamin D-, magnesium- and calcium deficiency.

ELIGIBILITY:
Inclusion Criteria:

* COPD-patients
* Unchanged medical treatment for COPD for the last 4 weeks
* Outpatients
* adults over 40 years

Exclusion Criteria:

* COPD exacerbation, which resulted in hospitalization and/or modification of medical treatment within 4 weeks
* Patients with other lung diseases, such as active tuberculosis, lung cancer, sarcoidosis and pulmonary fibrosis
* diseases affecting vitamin D and/or calcium and/or magnesium distribution
* Previous lung resection
* Treatment with systemic steroids
* Known addiction problems with alcohol and/or drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from the Department Of Resoiratory Diseases, Aarhus University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dahl, Professor, Study Director — Allergy Centre, Odense University Hospital; Sarah HA Hussein, MD, Principal Investigator — Department of Respiratory Diseases, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Publish as paper in Scientific journal

REFERENCES:
- [Derived] Hashim Ali Hussein S, Nielsen LP, Konow Bogebjerg Dolberg M, Dahl R. Serum magnesium and not vitamin D is associated with better QoL in COPD: A cross-sectional study. Respir Med. 2015 Jun;109(6):727-33. doi: 10.1016/j.rmed.2015.03.005. Epub 2015 Mar 27. PMID 25892292

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place in an outpatient clinic for respiratory diseases in Aarhus University Hospital, Denmark, during summertime in order to minimize seasonal variations of serum vitamin D.
Pre-assignment Details: Missed inclusion was due to either unstable disease (54 patients) or unwillingness to participate (87 patients).
Groups:
- Serum Vitamin D, Magnesium and Calcium Deficient Groups: Participants were distributed into wether they were serum vitamin D, magnesium and calcium sufficiency or deficiency.
Period: Overall Study
Arm/Group | Serum Vitamin D, Magnesium and Calcium Deficient Groups
Started | 143
Completed | 143
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Serum Vitamin D, Magnesium and Calcium Deficient Groups
Number analyzed (Participants) | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 99
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [63 to 74]
Gender [Count of Participants; unit: Participants]
  Female | 66
  Male | 77
Region of Enrollment [Number; unit: participants]
  Denmark | 143

OUTCOME MEASURES:

1. Primary Outcome: Serum Vitamin D
Description: vitamin D measured by p-25-hydroxy-vitamin D2 + D3, in mmol/L
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Serum Vitamin D: Participants' serum vitamin D
Arm/Group | Serum Vitamin D
Number analyzed (Participants) | 143
mmol/L | 75.13 (33.62)

2. Secondary Outcome: Lung Function Test
Description: Forced expiratory ventilation in 1 second, in percent of predicted
Time Frame: one year
Measure: Mean (Full Range); unit: percentage of predicted
Groups:
- Lung Function: lung function measured as forced expiratory volumes in 1 second.
Arm/Group | Lung Function
Number analyzed (Participants) | 143
percentage of predicted | 52 [33 to 71]

3. Secondary Outcome: Serum Magnesium
Description: Serum magnesium in plasma, in mmol/L
Time Frame: One year
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Serum Magnesium: Serum magnesium in plasma, in mmol/L
Arm/Group | Serum Magnesium
Number analyzed (Participants) | 143
mmol/L | 0.82 (0.08)

4. Secondary Outcome: Serum Calcium
Description: Serum ionized calcium, in mmol/L
Time Frame: One year
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Serum Calcium: Serum ionized calcium, in mmol/L
Arm/Group | Serum Calcium
Number analyzed (Participants) | 143
mmol/L | 1.23 (0.04)

5. Secondary Outcome: Quality of Life
Description: Quality of life measured by Chronic Obstructive Pulmonary Disease Assesment Test. Minimum score was 0 (no symptoms) and maximum score was 40 (many symptoms).
Time Frame: One year
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Quality of Life: Quality of life measured by Chronic Obstructive Pulmonary Disease Assesment Test
Arm/Group | Quality of Life
Number analyzed (Participants) | 143
units on a scale | 24 [22 to 28]

ADVERSE EVENTS:
Groups:
- EG000: Adverse Events were not collected for the 143 participants
Arm/Group | EG000
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The cross-sectional design. Some data (e.g. number of exacerbations past one year and smoking history) were self-reported and therefore, a risk of recall-bias cannot be excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes